CLINICAL TRIAL: NCT00414258
Title: The Holding Pilot Study: Feeding Analgesia in Preterm Infants
Brief Title: The Holding Study: Feeding Analgesia in Preterm Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Dr. Liisa Holsti, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C06 - 0347
Record Dates: First submitted 2006-12-19; First posted 2006-12-21 (Estimated); Last update posted 2011-04-14 (Estimated); Status verified 2011-04

CONDITIONS: Pain
Keywords: Pain Response
MeSH Terms: conditions — Pain | interventions — Lactation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: breastfeeding — See detailed description.

SUMMARY:
The purpose of this study is to compare the effects of mothers' skin-to-skin holding during feeding via a soother trainer with the effects of pacifier sucking on preterm infant biobehavioural responses during and immediately after a painful procedure

Hypothesis:

1. When held by their mothers during blood collection, preterm infants will show less pain reaction than when sucking on a pacifier.
2. Following holding during the blood collection, mothers will find no differences in their infants' feeding ability.

DETAILED DESCRIPTION:
Research Method:

In a between subjects, randomized design, 20 stable preterm infants born between 30-35 weeks gestational age will be studied. Infants will be randomized to one of two interventions which will take place during blood collections that are required for clinical management. For the standard care condition, infants will remain in their isolettes and will be positioned in prone and given a pacifier to suck on throughout the blood collection. For the holding condition, infants will be held skin-to-skin by their mothers and given breast milk using a soother trainer during the blood collection.

ELIGIBILITY:
Inclusion Criteria:

* Born between 30-35 weeks gestational age
* Mother has fluent English

Exclusion Criteria:

* CNS injury
* congenital anomaly
* active infection
* has had no surgeries or analgesics/sedatives in last 72 hours
* history of maternal drug exposure

Min Age: 3 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2006-09; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Videotaped and recorded at Baseline, Lance and Recovery:Neonatal Facial Coding System - total facial score; Heart Rate

SECONDARY OUTCOMES:
Videotaped and Recorded at Baseline, Lance and Recovery:Hand Movements; Sleep/Wake States
Samples taken at baseline and recovery;Salivary Cortisol sample

CONTACTS AND LOCATIONS:
Overall Officials: Liisa Holsti, Ph.D, Principal Investigator — University of British Columbia
Locations (1):
- Children's and Women's Health Centre of British Columbia, Special Care Nursery, Vancouver, British Columbia, Canada